CLINICAL TRIAL: NCT01015937
Title: Effect of Turmeric on Diabetic Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaheed Faghihi Hospital (Other)
Collaborators: Shiraz University of Medical Sciences (Other)
Responsible Party: Office of Vice Chancellor for research in Shiraz UMS, Shiraz University of Medical Science
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3997
Record Dates: First submitted 2009-11-16; First posted 2009-11-18 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2009-11

CONDITIONS: Diabetic Nephropathy; Proteinuria
Keywords: diabetes; nephropathy; turmeric; serum IL8; serum TGFb; serumINF; urinary IL8; urine TGFb
MeSH Terms: conditions — Diabetic Nephropathies; Proteinuria; Diabetes Mellitus; Kidney Diseases | interventions — turmeric extract; Curcumin; Dipeptidyl-Peptidases and Tripeptidyl-Peptidases; Receptor, Angiotensin, Type 1; Enalapril; Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Turmeric (Active Comparator): diabetic nephropathy patient
  more than 300 mg/proteinuria
  Interventions: Drug: Turmeric extract
- ACE inhibitor + ATI blocker (Active Comparator): diabetic nephropathy
  more than 300 mg/day proteinuria
  Interventions: Drug: Turmeric extract; Drug: Angiotensin-converting enzyme (ACE) inhibitor + Angiotensin-II type 1 receptor (ATI) blocker

INTERVENTIONS:
Drug: Turmeric extract — turmeric 500 mg TID for 45 days
  Other Names: turmeric
Drug: Angiotensin-converting enzyme (ACE) inhibitor + Angiotensin-II type 1 receptor (ATI) blocker — maximum dosage as patient tolerated for 45 days
  Other Names: enalapril; losartan
  Arms: ACE inhibitor + ATI blocker

SUMMARY:
The purpose of this study is to investigate whether turmeric is effective in improvement of diabetic nephropathy and in decrease in the amount of proteinuria and cytokine levels.

DETAILED DESCRIPTION:
Diabetic nephropathy is leading cause of ESRF that many therapy recommended for it. In this study, we investigate effect of turmeric on diabetic nephropathy, thus we selected diabetic nephropathy patients and divided them into 2 groups. One group received turmeric + ACE inhibitor + Angiotensin II receptor blocker (ARB) and the second group received only ACE inhibitor + ARB.

ELIGIBILITY:
Inclusion Criteria:

* diabetic nephropathy
* more than 300 mg proteinuria/day
* age more than 18 years old

Exclusion Criteria:

* DM type 1

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-03; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: maryam pakfetrat, assistant professor, Principal Investigator — Shiraz nephro-urology research center
Locations (1):
- Clinic, Shiraz, Fars, Iran